CLINICAL TRIAL: NCT06472232
Title: Efficacy and Safety of Chloroprocaine Versus Ropivacaine for Epidural Labor Analgesia Study: a Randomized, Double-blind, Controlled, Multicenter, Noninferiority Clinical Trial
Brief Title: Multicenter Study of Chloroprocaine Versus Ropivacaine for Epidural Labor Analgesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Beijing Obstetrics and Gynecology Hospital (Other); International Peace Maternity and Child Health Hospital (Other); Nanjing Medical University (Other); Anhui Women and Children's Medical Center (Unknown); Jiaxing Maternity and Child Health Care Hospital (Other); Gansu Maternal and Child Health Center (Unknown); Urumqi Maternal and Child Health Center (Unknown); Shengjing Hospital (Other); Zhongnan Hospital (Other); The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University (Unknown); Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-20240123-R
Record Dates: First submitted 2024-06-16; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Obstetric Labor
Keywords: labor analgesia; Chloroprocaine; Ropivacaine
MeSH Terms: interventions — chloroprocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroprocaine group (Experimental): Selection of local anesthetics for epidural labor analgesia with low concentration of chloroprocaine combined with sufentanil
  Interventions: Drug: Chloroprocaine
- Ropivacaine group (Placebo Comparator): Selection of local anesthetics for epidural labor analgesia with low concentration of ropivacaine combined with sufentanil
  Interventions: Drug: Chloroprocaine

INTERVENTIONS:
Drug: Chloroprocaine — Selection of low concentration of chloroprocaine as local anesthetic for labor analgesia
  Other Names: Ropivacaine

SUMMARY:
Women requiring epidural labor analgesia were randomized into two groups, one with the local anesthetic chloroprocaine and the other with ropivacaine. The primary outcome was to observe the analgesic scores of the two groups of drugs as well as adverse reactions.

DETAILED DESCRIPTION:
Mothers who met the study criteria vertebrae were included and then divided into two groups. Labor analgesia was provided by epidural anesthesia with a low concentration of local anesthetic (chloroprocaine or ropivacaine) combined with sufentanil. Data related to labor analgesia such as pain scores, motor tissue scores, and body temperature were collected and statistically analyzed to compare the efficacy and adverse effects of the two local anesthetics and to draw conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Primigravid women with full-term pregnancies scheduled for labor analgesia
* Determination of labor onset to cervical dilatation ≤ 5cm;
* Visual analogue scale (VAS) pain score during contractions >50 mm (0 mm = no pain at all, 100 mm = most intense pain);
* Age ≥20 years;
* American Society of Anesthesiologists (ASA) classification II
* Body mass index (BMI) between 18.5 and 30 kg/m2
* Height >155 cm
* Signed informed consent.

Exclusion Criteria:

* Twin or multiple pregnancies
* Hypertension
* Severe cardiopulmonary and hepatic or renal disease
* Severe pregnancy comorbidities such as preeclampsia, eclampsia, HELLP syndrome, placenta praevia, placental abruption, etc.
* Cephalopelvic disproportion
* History of allergy to local anesthesia
* Spinal deformity
* Contraindications to intrathecal anesthesia
* Refusal to participate in the stud

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2024-06-18 (Estimated); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of effective analgesia | 30 min after the first epidural addition at the beginning of labor analgesia
  Percentage of effective analgesia within 30 min after the first epidural addition at the beginning of labor analgesia in both groups